CLINICAL TRIAL: NCT06345976
Title: Functional Impairment in Albinism
Acronym: PLAIB
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RLX_2023_10
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Albinism, Ocular
MeSH Terms: conditions — Albinism, Ocular | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: questionnaire — On-line self-questionnaire, in the form of an 18-question form, the link to which is sent by e-mail to patients with albinism who have agreed to take part in the study.

SUMMARY:
Albinism is a genetic and hereditary anomaly that affects pigmentation. This pathology is characterized by a deficit in melanin production. In humans, the clinical diagnosis of albinism is based on a number of factors, including :

* In the integumentary region: fair skin tone, with white hair, eyelashes and eyebrows.
* Ophthalmological: reduced visual acuity, photophobia, nystagmus, transilluminated blue irises, hypopigmentation of the retina at the back of the eye with fovea plana.

As treatment options begin to emerge for certain albinism-induced anomalies (including, for example, the depigmentation that causes photophobia), it is desirable to understand what these patients' complaints are, and to gather their views on the emergence of treatments targeting just one of their complaints, namely glare.

ELIGIBILITY:
Inclusion Criteria:

* All patients with albinism
* Patients > 18 years of age
* Non-opposition to study participation

Exclusion Criteria:

No diagnosis according to Kruijt et al. criteria Impossibility (visual, technological) of completing questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified in the hospital's database, or may be contacted by patient associations.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
To determine whether patients with albinism would be interested in a treatment that could improve their glare without improving their visual acuity. | Day0
  To determine whether patients with albinism would be interested in a treatment that could improve their glare without improving their visual acuity.
  Percentage of positive responses to question "Would you be interested in the possibility of a treatment for glare if it did not improve the quality of vision or visual stability?"

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation A. de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No